CLINICAL TRIAL: NCT01507987
Title: St.Jude Medical Cardiac Lead Assessment Study
Acronym: CLAS
Status: Completed | Type: Observational
Sponsor: Abbott Medical Devices (Industry)
Responsible Party: Sponsor
Other Study IDs: 60039775/K; CRD-619 (Other: St. Jude Medical)
Record Dates: First submitted 2012-01-06; First posted 2012-01-11 (Estimated); Results first posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-07

CONDITIONS: Externalized Conductors; Visual Lead Anomalies; Electrical Dysfunction
Keywords: Externalized Conductors, visual lead an

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with SJM leads implanted: Patient has at least one market released Riata, Riata ST, QuickSite/QuickFlex, or Durata lead implanted
  Interventions: Device: Implanted with one or more of the following SJM leads: Riata leads, RiataST leads, Durata leads, and QuickSite/QuickFlex leads

INTERVENTIONS:
Device: Implanted with one or more of the following SJM leads: Riata leads, RiataST leads, Durata leads, and QuickSite/QuickFlex leads — Riata leads implanted between 2002-2009 Riata ST leads implanted between 2006-2009 Quicksite or QuickFlex leads implanted between 2006-2010 Durata leads implanted between 2008-2010
  Subjects were followed for three years and cinefluoroscopy imaging was done annually to determine prevalence of externalized conductors or other visual lead anomalies

SUMMARY:
The Cardiac Lead Assessment Study (CLAS) is designed as a prospective, non-randomized, multi-center, international postmarket surveillance study under 522 Order PS120111 (August 16, 2012).

DETAILED DESCRIPTION:
The objective of this study was to determine the prevalence and incidence of externalized conductors and other visual lead anomalies (as evidenced by imaging) and the risk of progression to electrical dysfunction in subjects with one or more of the following St. Jude Medical (SJM) cardiac leads: Riata leads, Riata ST leads, Durata and/or QuickSite/QuickFlex Cardiac Resynchronization Therapy (CRT) leads.

ELIGIBILITY:
Inclusion Criteria:

1. Patient has a market released SJM Implantable Cardioverter Defibrillator (ICD), CRT-D or CRT-P already implanted.
2. Patient has at least one market released Riata/ Riata ST/QuickSite/QuickFlex/Durata already implanted in which the lead model number and lead implant date is indicated in Table 1 (see protocol attached.)
3. Have the ability to provide informed consent for study participation and be willing to comply with the prescribed evaluations as detailed in this study plan.
4. Are 18 years or above

Exclusion Criteria:

1. Patient is currently pregnant.
2. Enrolled or intend to participate in a clinical drug and/or device study, which could confound the results of this trial as determined by SJM, during the course of this clinical study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients that have a market released St. Jude Medical Implantable Cardioverter Defibrillator (ICD) or Cardiac Resynchronization Therapy - Defibrillator (CRT-D) already implanted and also have at least one market released Riata/ Riata ST/QuickSite/QuickFlex/Durata already implanted.
Sampling Method: Probability Sample
Enrollment: 2216 (Actual)
Dates: Start 2013-03 (Actual); Primary Completion 2019-06 (Actual); Study Completion 2019-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (45):
- United States (41):
  - Cardiology, P.C., Birmingham, Alabama
  - University Hospital of Alabama at Birmingham, Birmingham, Alabama
  - Heart Center Research, Huntsville, Alabama
  - Arizona Arrhythmia Consultants, Scottsdale, Arizona
  - Arkansas Heart Hospital, Little Rock, Arkansas
  - Scripps Green Hospital, La Jolla, California
  - Kaiser Permanente Los Angeles Medical Center, Los Angeles, California
  - Cardiac Rhythm Specialists, Reseda, California
  - Mercy Medical Group, Sacramento, California
  - St. Joseph's Medical Center, Stockton, California
  - Penrose St. Francis Health Services, Colorado Springs, Colorado
  - Naples Heart Rhytm Specialists, PA, Naples, Florida
  - Redmond Regional Medical Center, Rome, Georgia
  - OSF Healthcare Cardiovascular Institute, Peoria, Illinois
  - Mid-America Cardiology Associates, PC, Kansas City, Kansas
  - Heart Clinic of Hammond, LLC, Hammond, Louisiana
  - Ochsner Medical Center, New Orleans, Louisiana
  - Massachusetts General Hospital, Boston, Massachusetts
  - Sparrow Clinical Research Institute, Lansing, Michigan
  - Jackson Heart Clinic, Jackson, Mississippi
  - Cardiology Associates of North Mississippi, Tupelo, Mississippi
  - Methodist Physicians Clinic-Heart Consultants, Omaha, Nebraska
  - Deborah Heart and Lung, Browns Mills, New Jersey
  - New Mexico Heart Institute, Albuquerque, New Mexico
  - Asheville Cardiology Associates, Asheville, North Carolina
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio State University, Columbus, Ohio
  - The Toledo Hospital, Toledo, Ohio
  - Providence Heart & Vascular Institute, Portland, Oregon
  - Saint Vincent Consultants in Cardiovascular Diseases, Erie, Pennsylvania
  - Drexel University College oF Medicine, Philadelphia, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Donald Guthrie Foundation for Education and Research, Sayre, Pennsylvania
  - Wellspan Health, York, Pennsylvania
  - Sutherland Cardiology Clinic, Germantown, Tennessee
  - Mountain States Medical Group Cardiology, Johnson City, Tennessee
  - Arrhythmia Consultants, Memphis, Tennessee
  - South Texas Cardiovascular Consultants, San Antonio, Texas
  - University of Utah Hospital, Salt Lake City, Utah
  - Sentara Norfolk General Hospital, Norfolk, Virginia
  - Aurora Medical Group, Milwaukee, Wisconsin
- QE II Health Sciences, Halifax, Nova Scotia, Canada
- Japan (3):
  - University of Tsukuba Hospital, Tsukuba, Ibaraki
  - Osaka City University Hospital, Osaka, Osaka
  - Kyoto-Katsura Hospital, Kyoto

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study enrolled a total of 2,216 subjects at 45 sites to achieve an evaluable sample size of at least 1,401 subjects. The first subject enrolled in this study on March 20, 2013 and enrollment was completed in June, 2016 with the last follow-up completed in June 13 2019.
Pre-assignment Details: A subject that has at least one market released lead implanted was eligible for enrollment in the study. Subjects could have more than one study lead implanted. Each lead group was considered separately for independent analyses.
Units Other Than Participants: implants
Groups:
- Durata Leads: Durata leads implanted between 2008-2010
- Riata Leads: Riata leads implanted between 2002-2009
- Riata ST: Riata ST leads implanted 2006-2009
- QuickSite/QuickFlex: QuickSite/QuickFlex implanted 2006-2010
Period: Overall Study
Arm/Group | Durata Leads | Riata Leads | Riata ST | QuickSite/QuickFlex
Started | 982; 982 implants | 670; 670 implants | 458; 458 implants | 737; 737 implants
Completed | 618; 618 implants | 335; 335 implants | 252; 252 implants | 480; 480 implants
Not Completed | 364; 364 implants | 335; 335 implants | 206; 206 implants | 257; 257 implants

BASELINE CHARACTERISTICS:
Population: The study enrolled a total of 2,216 study participants
Groups:
- All Subjects Enrolled in the Study: Demographics for all enrolled patients (N=2216)
Arm/Group | All Subjects Enrolled in the Study
Number analyzed (Participants) | 2216
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 600
  Male | 1616
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 56
  Not Hispanic or Latino | 2158
  Unknown or Not Reported | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 8
  Asian | 91
  Native Hawaiian or Other Pacific Islander | 3
  Black or African American | 335
  White | 1770
  More than one race | 0
  Unknown or Not Reported | 9
Region of Enrollment [Number; unit: participants]
  Canada | 48
  United States | 2085
  Japan | 83

OUTCOME MEASURES:

1. Primary Outcome: Number of Leads With Electrical Dysfunction
Description: The prevalence of electrical dysfunction was calculated as the number of leads that have electrical dysfunction through three years of follow-up for the 4 lead groups divided by total number of leads in enrolled patients in each of the 4 lead groups.
Time Frame: This outcome is assessed at enrollment and over the course of 3 years of follow-up
Population: All SJM leads enrolled in the study with Durata, Riata, Riata ST, or QuickSite/QuickFlex leads
Measure: Count of Units; unit: implanted leads
Units Other Than Participants: implanted leads
Arm/Group | Durata Leads | Riata Leads | Riata ST | QuickSite/QuickFlex
Number analyzed (Participants) | 982 | 670 | 458 | 737
Number analyzed (implanted leads) | 982 | 670 | 458 | 737
implanted leads | 24 | 27 | 15 | 2

2. Primary Outcome: Number of Leads With Externalized Conductors
Description: The prevalence of externalized conductors was calculated as the number of leads that have been shown to have externalized conductors by imaging at the time of enrollment in each of the 4 lead groups divided by total number of leads in enrolled patients in each of the 4 lead groups
Time Frame: This outcome is assessed at enrollment
Population: All SJM leads enrolled in the study with Durata, Riata, Riata ST, or QuickSite/QuickFlex leads
Measure: Count of Units; unit: implanted leads
Units Other Than Participants: implanted leads
Arm/Group | Durata Leads | Riata Leads | Riata ST | QuickSite/QuickFlex
Number analyzed (Participants) | 973 | 660 | 452 | 723
Number analyzed (implanted leads) | 973 | 660 | 452 | 723
implanted leads | 0 | 144 | 44 | 10

3. Primary Outcome: Number of Other Visual Lead Anomalies by Each Subcategory (Fracture, Kink, Subclavian Crush, Other Irregularities)
Description: The prevalence of other visual lead anomalies (by each subcategory) was calculated as the number of leads that have been shown to have other visual anomaly (by each subcategory) at the time of enrollment in each of the 4 lead groups divided by total number of leads in enrolled patients in each of the 4 lead groups.
Time Frame: This outcome is assessed at enrollment
Measure: Count of Units; unit: implanted leads
Units Other Than Participants: implanted leads
Arm/Group | Durata Leads | Riata Leads | Riata ST | QuickSite/QuickFlex
Number analyzed (Participants) | 974 | 646 | 454 | 724
Number analyzed (implanted leads) | 974 | 646 | 454 | 724
implanted leads | 7 | 19 | 7 | 4

4. Primary Outcome: The Annual Hazard Rate of Lead Electrical Dysfunction in the Riata, Riata ST, QuickSite/QuickFlex (1056T, 1058T, 1156T, 1158T) and Durata Leads.
Description: Annual hazard rate is the proportion of number of leads with electrical dysfunction to the total number of lead follow-up years.
Time Frame: This outcome is assessed from enrollment through the course of 3 years of follow-up
Population: The annual hazard rate was assessed separately in each of the 4 lead groups.
Measure: Number; unit: leads with electrical dysfunction/years
Units Other Than Participants: implanted leads
Arm/Group | Durata Leads | Riata Leads | Riata ST | QuickSite/QuickFlex
Number analyzed (Participants) | 982 | 670 | 458 | 737
Number analyzed (implanted leads) | 982 | 670 | 458 | 737
leads with electrical dysfunction/years | 0.010 | 0.019 | 0.014 | 0.001

5. Primary Outcome: The Annual Hazard Rate of New Cases of Externalized Conductors (From Enrollment to Year 1) in the Riata, Riata ST, QuickSite/QuickFlex (1056T, 1058T, 1156T, 1158T) and Durata Leads.
Description: Annual hazard rate calculated as ratio of all leads that are adjudicated by the committee and a have definite outcome of presence of externalized conductors to total follow-up years from enrollment to year 1
Time Frame: year 1 follow-up
Population: The annual hazard rate was assessed separately in each of the 4 lead groups.
Measure: Number (95% Confidence Interval); unit: leads with externalized conductors/years
Units Other Than Participants: implanted leads
Arm/Group | Durata Leads | Riata Leads | Riata ST | QuickSite/QuickFlex
Number analyzed (Participants) | 808 | 375 | 316 | 556
Number analyzed (implanted leads) | 808 | 375 | 316 | 556
leads with externalized conductors/years | 0.0025 [0.0003 to 0.0089] | 0.0480 [.0287 to 0.0748] | 0.0158 [0.0052 to 0.0365] | 0.0288 [0.0165 to 0.0463]

6. Primary Outcome: The Annual Hazard Rate of New Cases of Externalized Conductors (From Year 1 to Year 2) in the Riata, Riata ST, QuickSite/QuickFlex (1056T, 1058T, 1156T, 1158T) and Durata Leads.
Description: Annual hazard rate calculated as ratio of all leads that are adjudicated by the committee and a have definite outcome of presence of externalized conductors to total follow-up years from year 1 to year 2
Time Frame: year 1 to year 2 follow-up
Population: The annual hazard rate was assessed separately in each of the 4 lead groups.
Measure: Number (95% Confidence Interval); unit: leads with externalized conductors/years
Units Other Than Participants: implanted leads
Arm/Group | Durata Leads | Riata Leads | Riata ST | QuickSite/QuickFlex
Number analyzed (Participants) | 687 | 301 | 256 | 462
Number analyzed (implanted leads) | 687 | 301 | 256 | 462
leads with externalized conductors/years | 0.0015 [0 to 0.0081] | 0.0897 [0.0599 to 0.1278] | 0.0234 [0.0086 to 0.0503] | 0.0087 [0.0024 to 0.022]

7. Primary Outcome: The Annual Hazard Rate of New Cases of Externalized Conductors (From Year 2 to Year 3) in the Riata, Riata ST, QuickSite/QuickFlex (1056T, 1058T, 1156T, 1158T) and Durata Leads.
Description: Annual hazard rate calculated as ratio of all leads that are adjudicated by the committee and a have definite outcome of presence of externalized conductors to total follow-up years from year 2 to year 3
Time Frame: year 2 to year 3 follow-up
Population: The annual hazard rate was assessed separately in each of the 4 lead groups.
Measure: Number (95% Confidence Interval); unit: leads with externalized conductors/years
Units Other Than Participants: implanted leads
Arm/Group | Durata Leads | Riata Leads | Riata ST | QuickSite/QuickFlex
Number analyzed (Participants) | 570 | 228 | 206 | 362
Number analyzed (implanted leads) | 570 | 228 | 206 | 362
leads with externalized conductors/years | 0.0035 [0.0004 to 0.0126] | 0.0658 [0.0373 to 0.1062] | 0.0097 [0.0012 to 0.0346] | 0.0110 [0.003 to 0.0280]

8. Primary Outcome: The Annual Hazard Rate of New Cases of Other Visual Lead Anomalies by Each Subcategory (From Enrollment to Year 1) in the Riata, Riata ST, QuickSite/QuickFlex (1056T, 1058T, 1156T, 1158T) and Durata Leads
Description: Annual hazard rate calculated as proportion of leads adjudicated by the committee and a have definite outcome of presence of other visual lead anomaly to total follow up years from enrollment to year 1
Time Frame: This outcome is assessed from enrollment to year 1
Population: The annual hazard rate was assessed separately in each of the 4 lead groups.
Measure: Number (95% Confidence Interval); unit: leads w other visual lead anomaly/years
Units Other Than Participants: implanted leads
Arm/Group | Durata Leads | Riata Leads | Riata ST | QuickSite/QuickFlex
Number analyzed (Participants) | 803 | 461 | 343 | 571
Number analyzed (implanted leads) | 803 | 461 | 343 | 571
leads w other visual lead anomaly/years | 0.0025 [0.0003 to 0.0090] | 0.0108 [0.0035 to 0.0251] | 0.0117 [0.0032 to 0.0296] | 0.0053 [0.0011 to 0.0153]

9. Primary Outcome: The Annual Hazard Rate of New Cases of Other Visual Lead Anomalies by Each Subcategory (From Year 1 to Year 2) in the Riata, Riata ST, QuickSite/QuickFlex (1056T, 1058T, 1156T, 1158T) and Durata Leads
Description: Annual hazard rate calculated as proportion of leads adjudicated by the committee and a have definite outcome of presence of other visual lead anomaly to total follow up years from year 1 to year 2
Time Frame: This outcome is assessed from year 1 to year 2 of follow-up
Population: The annual hazard rate was assessed separately in each of the 4 lead groups.
Measure: Number (95% Confidence Interval); unit: leads w other visual lead anomaly/years
Units Other Than Participants: implanted leads
Arm/Group | Durata Leads | Riata Leads | Riata ST | QuickSite/QuickFlex
Number analyzed (Participants) | 254 | 374 | 286 | 482
Number analyzed (implanted leads) | 254 | 374 | 286 | 482
leads w other visual lead anomaly/years | 0 [0 to 0.0054] | 0.0027 [0.0001 to 0.0148] | 0.0070 [0.0008 to 0.025] | 0.0021 [0.0001 to 0.0115]

10. Primary Outcome: The Annual Hazard Rate of New Cases of Other Visual Lead Anomalies by Each Subcategory (From Year 2 to Year 3) in the Riata, Riata ST, QuickSite/QuickFlex (1056T, 1058T, 1156T, 1158T) and Durata Leads
Description: Annual hazard rate calculated as proportion of leads adjudicated by the committee and a have definite outcome of presence of other visual lead anomaly to total follow up years from year 2 to year 3
Time Frame: This outcome is assessed from year 2 to year 3 follow-up
Population: The annual hazard rate was assessed separately in each of the 4 lead groups.
Measure: Number (95% Confidence Interval); unit: leads w other visual lead anomaly/years
Units Other Than Participants: implanted leads
Arm/Group | Durata Leads | Riata Leads | Riata ST | QuickSite/QuickFlex
Number analyzed (Participants) | 565 | 305 | 229 | 387
Number analyzed (implanted leads) | 565 | 305 | 229 | 387
leads w other visual lead anomaly/years | 0 [0 to 0.0065] | 0.0066 [0.0008 to 0.0235] | 0 [0 to 0.0160] | 0 [0 to 0.0095]

11. Secondary Outcome: Estimation of Cumulative Lead Anomaly Events From Time of Detecting Externalized Conductors to Electrical Dysfunction, by Year of Initial Implant
Description: Kaplan-Meier analysis of time from externalized conductors (EC) to electrical dysfunction, by year of initial implant. Count of cumulative lead anomaly events from time of detecting EC
Time Frame: This outcome is assessed from time of detecting EC till the course of 3 years of follow-up
Population: N at risk from detecting externalized conductors at each follow-up time point
Measure: Number; unit: lead anomaly events
Units Other Than Participants: Implant Leads
Groups:
- Durata Leads Lead Age: Less Than 4 Years: lead age: less than 4 years
- Durata Leads Lead Age: 4 to Less Than 5 Years: lead age: 4 to less than 5 years
- Durata Leads Lead Age: 5 Years or Greater: lead age: 5 years or greater
- Riata Leads Lead Age: Less Than 6 Years: lead age: less than 6 years
- Riata Leads Lead Age: 6-less Than 7 Years: lead age: 6-less than 7 years
- Riata Leads Lead Age: 7 Years or Greater: lead age: 7 years or greater
- Riata ST Lead Age: Less Than 5.5 Years: lead age: less than 5.5 years
- Riata ST Leads Lead Age: Greater Than or Equal to 5.5 Years: lead age: greater than or equal to 5.5 years
- QuickSite/QuickFlex Lead Age: Less Than 5 Years: lead age: less than 5 years
- QuickSite/QuickFlex Leads Lead Age: 5 to Less Than 6 Years: lead age: 5 to less than 6 years
- QuickSite/QuickFlex Leads Lead Age: Greater Than or Equal to 6 Years: lead age: greater than or equal to 6 years
Arm/Group | Durata Leads Lead Age: Less Than 4 Years | Durata Leads Lead Age: 4 to Less Than 5 Years | Durata Leads Lead Age: 5 Years or Greater | Riata Leads Lead Age: Less Than 6 Years | Riata Leads Lead Age: 6-less Than 7 Years | Riata Leads Lead Age: 7 Years or Greater | Riata ST Lead Age: Less Than 5.5 Years | Riata ST Leads Lead Age: Greater Than or Equal to 5.5 Years | QuickSite/QuickFlex Lead Age: Less Than 5 Years | QuickSite/QuickFlex Leads Lead Age: 5 to Less Than 6 Years | QuickSite/QuickFlex Leads Lead Age: Greater Than or Equal to 6 Years
Number analyzed (Participants) | 1 | 2 | 2 | 42 | 67 | 93 | 23 | 34 | 12 | 12 | 15
Number analyzed (Implant Leads) | 1 | 2 | 2 | 42 | 67 | 93 | 23 | 34 | 12 | 12 | 15
lead anomaly events
  year 0 from detecting externalized conductor | 0 | 0 | 0 | 1 | 1 | 3 | 0 | 1 | 0 | 0 | 0
  year 1 from detecting externalized conductor: number analyzed (Participants) | 1 | 2 | 2 | 30 | 43 | 63 | 16 | 26 | 11 | 9 | 13
  year 1 from detecting externalized conductor: number analyzed (Implant Leads) | 1 | 2 | 2 | 30 | 43 | 63 | 16 | 26 | 11 | 9 | 13
  year 1 from detecting externalized conductor | 0 | NA — no data available | NA — no data available | 2 | 1 | 5 | 0 | 2 | 0 | 0 | 0
  year 2 from detecting externalized conductor: number analyzed (Participants) | 1 | 2 | 2 | 19 | 27 | 38 | 8 | 22 | 5 | 6 | 9
  year 2 from detecting externalized conductor: number analyzed (Implant Leads) | 1 | 2 | 2 | 19 | 27 | 38 | 8 | 22 | 5 | 6 | 9
  year 2 from detecting externalized conductor | NA — no data available | NA — no data available | NA — no data available | 2 | 2 | 6 | 1 | 2 | 0 | 0 | 0
  year 3 from detecting externalized conductor: number analyzed (Participants) | 1 | 2 | 2 | 8 | 12 | 15 | 5 | 8 | 5 | 1 | 5
  year 3 from detecting externalized conductor: number analyzed (Implant Leads) | 1 | 2 | 2 | 8 | 12 | 15 | 5 | 8 | 5 | 1 | 5
  year 3 from detecting externalized conductor | NA — no data available | NA — no data available | NA — no data available | 2 | 3 | 6 | 1 | 4 | NA — no data available | 0 | 0

12. Secondary Outcome: Estimation of Cumulative Lead Anomaly Events From Time of Detecting Other Visual Lead Anomaly to Electrical Dysfunction, by Year of Initial Implant
Description: Kaplan-Meier analysis of time from other visual lead anomaly to electrical dysfunction, by year of initial implant. Count of cumulative lead anomaly events from time of detecting other visual lead anomaly
Time Frame: This outcome is assessed from time of detecting other visual lead anomaly till the course of 3 years of follow-up
Population: N at risk from detecting other visual lead anomaly
Measure: Number; unit: lead anomaly events
Units Other Than Participants: Implant Leads
Arm/Group | Durata Leads Lead Age: Less Than 4 Years | Durata Leads Lead Age: 4 to Less Than 5 Years | Durata Leads Lead Age: 5 Years or Greater | Riata Leads Lead Age: Less Than 6 Years | Riata Leads Lead Age: 6-less Than 7 Years | Riata Leads Lead Age: 7 Years or Greater | Riata ST Lead Age: Less Than 5.5 Years | Riata ST Leads Lead Age: Greater Than or Equal to 5.5 Years | QuickSite/QuickFlex Lead Age: Less Than 5 Years | QuickSite/QuickFlex Leads Lead Age: 5 to Less Than 6 Years | QuickSite/QuickFlex Leads Lead Age: Greater Than or Equal to 6 Years
Number analyzed (Participants) | 5 | 2 | 2 | 7 | 10 | 10 | 6 | 7 | 2 | 3 | 3
Number analyzed (Implant Leads) | 5 | 2 | 2 | 7 | 10 | 10 | 6 | 7 | 2 | 3 | 3
lead anomaly events
  0 years follow up from detecting other visual lead anomaly | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  1 years follow up from detecting other visual lead anomaly: number analyzed (Participants) | 4 | 2 | 2 | 5 | 8 | 7 | 5 | 5 | 2 | 3 | 2
  1 years follow up from detecting other visual lead anomaly: number analyzed (Implant Leads) | 4 | 2 | 2 | 5 | 8 | 7 | 5 | 5 | 2 | 3 | 2
  1 years follow up from detecting other visual lead anomaly | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  2 years follow up from detecting other visual lead anomaly: number analyzed (Participants) | 2 | 2 | 2 | 3 | 6 | 4 | 2 | 3 | 1 | 3 | 1
  2 years follow up from detecting other visual lead anomaly: number analyzed (Implant Leads) | 2 | 2 | 2 | 3 | 6 | 4 | 2 | 3 | 1 | 3 | 1
  2 years follow up from detecting other visual lead anomaly | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  3 years follow up from detecting other visual lead anomaly: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 3 | 1 | 1 | 1
  3 years follow up from detecting other visual lead anomaly: number analyzed (Implant Leads) | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 3 | 1 | 1 | 1
  3 years follow up from detecting other visual lead anomaly | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Number of Participants With an Adverse Event Through 30 Days Post-intervention for Lead (e.g. Extraction, Abandonment, Revision, Other).
Description: Number of participants with adverse events within 30 days associated with study lead related interventions for each lead group
Time Frame: within 30 days associated with study lead related interventions
Population: Subject has at least one market released Riata, Riata ST, QuickSite/QuickFlex, or Durata lead implanted
Measure: Count of Participants; unit: Participants
Groups:
- Riata ST Leads: Riata ST leads implanted between 2006-2009
- QuickSite/QuickFlex Leads: Quicksite or QuickFlex leads implanted between 2006-2010
Arm/Group | Durata Leads | Riata Leads | Riata ST Leads | QuickSite/QuickFlex Leads
Number analyzed (Participants) | 982 | 670 | 458 | 737
Participants
  Lead dislodgement or migration | 1 | 0 | 0 | 0
  lead insulation damage | 0 | 0 | 0 | 1
  phrenic nerve/diaphragmatic stimulation | 0 | 0 | 0 | 1

14. Secondary Outcome: Estimation of Cumulative Lead Anomaly Events From Time of Detecting Externalized Conductors to Clinical Intervention, by Year of Initial Implant
Description: time from externalized conductors to clinical intervention for all lead subgroups.
Time Frame: This outcome is assessed from time of detection of externalized conductor to 3 years follow-up
Population: N at risk from time of externalized conductors at each follow-up period
Measure: Number; unit: lead anomaly events
Units Other Than Participants: Implant Leads
Arm/Group | Durata Leads Lead Age: Less Than 4 Years | Durata Leads Lead Age: 4 to Less Than 5 Years | Durata Leads Lead Age: 5 Years or Greater | Riata Leads Lead Age: Less Than 6 Years | Riata Leads Lead Age: 6-less Than 7 Years | Riata Leads Lead Age: 7 Years or Greater | Riata ST Lead Age: Less Than 5.5 Years | Riata ST Leads Lead Age: Greater Than or Equal to 5.5 Years | QuickSite/QuickFlex Lead Age: Less Than 5 Years | QuickSite/QuickFlex Leads Lead Age: 5 to Less Than 6 Years | QuickSite/QuickFlex Leads Lead Age: Greater Than or Equal to 6 Years
Number analyzed (Participants) | 1 | 2 | 2 | 42 | 67 | 93 | 23 | 34 | 12 | 12 | 15
Number analyzed (Implant Leads) | 1 | 2 | 2 | 42 | 67 | 93 | 23 | 34 | 12 | 12 | 15
lead anomaly events
  0 years from detecting EC | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
  1 year from detecting EC: number analyzed (Participants) | 1 | 2 | 2 | 31 | 43 | 63 | 16 | 26 | 11 | 9 | 13
  1 year from detecting EC: number analyzed (Implant Leads) | 1 | 2 | 2 | 31 | 43 | 63 | 16 | 26 | 11 | 9 | 13
  1 year from detecting EC | 0 | 1 | 1 | 2 | 5 | 11 | 3 | 4 | 0 | 0 | 0
  2 years from detecting EC: number analyzed (Participants) | 1 | 2 | 2 | 19 | 27 | 38 | 8 | 22 | 5 | 6 | 9
  2 years from detecting EC: number analyzed (Implant Leads) | 1 | 2 | 2 | 19 | 27 | 38 | 8 | 22 | 5 | 6 | 9
  2 years from detecting EC | NA — no data available | 1 | 1 | 3 | 7 | 15 | 6 | 4 | 1 | 0 | 0
  3 years from detecting EC: number analyzed (Participants) | 1 | 2 | 2 | 8 | 12 | 38 | 8 | 8 | 5 | 1 | 5
  3 years from detecting EC: number analyzed (Implant Leads) | 1 | 2 | 2 | 8 | 12 | 38 | 8 | 8 | 5 | 1 | 5
  3 years from detecting EC | NA — no data available | 1 | 1 | 4 | 8 | 18 | 6 | 6 | 1 | 0 | 0

15. Secondary Outcome: Estimation of Lead Anomaly Events From Time of Other Visual Lead Anomalies by Each Subcategory to Clinical Intervention, by Year of Initial Implant
Description: Kaplan-Meier analysis of time from visual lead anomalies for all lead and lead age subcategories to clinical intervention
Time Frame: This outcome is assessed from time of detection of other visual lead anomaly until 3 years of follow-up
Population: N at risk from time of detecting visual lead anomaly at each follow-up period
Measure: Number; unit: lead anomaly events
Units Other Than Participants: Implant Leads
Arm/Group | Durata Leads Lead Age: Less Than 4 Years | Durata Leads Lead Age: 4 to Less Than 5 Years | Durata Leads Lead Age: 5 Years or Greater | Riata Leads Lead Age: Less Than 6 Years | Riata Leads Lead Age: 6-less Than 7 Years | Riata Leads Lead Age: 7 Years or Greater | Riata ST Lead Age: Less Than 5.5 Years | Riata ST Leads Lead Age: Greater Than or Equal to 5.5 Years | QuickSite/QuickFlex Lead Age: Less Than 5 Years | QuickSite/QuickFlex Leads Lead Age: 5 to Less Than 6 Years | QuickSite/QuickFlex Leads Lead Age: Greater Than or Equal to 6 Years
Number analyzed (Participants) | 5 | 2 | 2 | 7 | 10 | 10 | 6 | 7 | 2 | 3 | 3
Number analyzed (Implant Leads) | 5 | 2 | 2 | 7 | 10 | 10 | 6 | 7 | 2 | 3 | 3
lead anomaly events
  0 years from detection other visual lead anomaly | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  1 years from detection other visual lead anomaly: number analyzed (Participants) | 4 | 2 | 2 | 5 | 8 | 7 | 5 | 5 | 2 | 3 | 2
  1 years from detection other visual lead anomaly: number analyzed (Implant Leads) | 4 | 2 | 2 | 5 | 8 | 7 | 5 | 5 | 2 | 3 | 2
  1 years from detection other visual lead anomaly | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
  2 years from detection other visual lead anomaly: number analyzed (Participants) | 2 | 2 | 2 | 3 | 6 | 4 | 2 | 3 | 1 | 3 | 1
  2 years from detection other visual lead anomaly: number analyzed (Implant Leads) | 2 | 2 | 2 | 3 | 6 | 4 | 2 | 3 | 1 | 3 | 1
  2 years from detection other visual lead anomaly | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0
  3 years from detection other visual lead anomaly: number analyzed (Participants) | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 3 | 1 | 1 | 1
  3 years from detection other visual lead anomaly: number analyzed (Implant Leads) | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 3 | 1 | 1 | 1
  3 years from detection other visual lead anomaly | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 0

16. Secondary Outcome: Comparison of Number of Patients With Externalized Conductors to Number of Patients Without Externalized Conductors (EC)
Description: Comparison of patients with EC to those without EC: lead size effect on number of patients with or without EC (7F and 8F are lead sizes, F = French). Riata leads have 8F diameter and Riata ST leads have 7F diameter. The Riata/Riata ST families of leads were used for this comparison only to determine whether the difference in lead size (with the silicon material and other lead design factors controlled for) had an effect on externalization of conductors.
Time Frame: This outcome is assessed from enrollment till the course of 3 years of follow-up
Population: Patients with Riata or Riata ST leads.
Measure: Count of Participants; unit: Participants
Groups:
- With Externalized Conductors (EC): EC identified
- Without Externalized Conductors (EC): No EC identified
Arm/Group | With Externalized Conductors (EC) | Without Externalized Conductors (EC)
Number analyzed (Participants) | 261 | 851
Participants
  7F lead size (Riata ST) | 57 | 395
  8F lead size (Riata) | 204 | 456

17. Secondary Outcome: Comparison of Patients With Electrical Dysfunction to Those Without Electrical Dysfunction (ED).
Description: Comparison of patients with ED to those without ED: subject age effect on ED
Time Frame: This outcome is assessed from enrollment till the course of 3 years of follow-up
Population: Patients implanted with SJM Riata, Riata ST, Durata, or QuickSite/QuickFlex leads. Leads were combined for this analysis to compare patient groups with and without electrical dysfunction based on age (irrespective of lead implant type)
Measure: Mean (Standard Deviation); unit: years
Groups:
- With Electrical Dysfunction (ED): ED identified
- Without Electrical Dysfunction (ED): No ED identified
Arm/Group | With Electrical Dysfunction (ED) | Without Electrical Dysfunction (ED)
Number analyzed (Participants) | 68 | 2148
years | 61.8 (13.4) | 67.2 (11.9)

ADVERSE EVENTS:
Time Frame: From enrollment to 3 years of follow-up period
Groups:
- Durata Leads: Subjects implanted with SJM Durata leads
- Riata Leads: Subjects implanted with Riata leads
- Riata ST Leads: Subjects implanted with Riata ST leads
- QuickSite/QuickFlex Leads: Subjects implanted with QuickSite/QuickFlex leads
Arm/Group | Durata Leads | Riata Leads | Riata ST Leads | QuickSite/QuickFlex Leads
All-Cause Mortality (participants affected / at risk) | 130/982 | 111/670 | 64/458 | 135/737
Serious Adverse Events (participants affected / at risk) | 26/982 | 28/670 | 22/458 | 7/737
Other Adverse Events (participants affected / at risk) | 20/982 | 14/670 | 9/458 | 11/737
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durata Leads (N=982) | Riata Leads (N=670) | Riata ST Leads (N=458) | QuickSite/QuickFlex Leads (N=737)
Abnormal high voltage lead impredance (Product Issues) | 3 (3) | 5 (5) | 5 (5) | 0 (0)
Abnormal Pacing Impedance (Product Issues) | 8 (8) | 2 (2) | 0 (0) | 0 (0)
Decline in R Wave Sensing (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated pacing thresholds (Product Issues) | 0 (0) | 4 (4) | 1 (1) | 2 (2)
Externalized Conductor (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lead dislodgement or migration (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
lead fracture (Product Issues) | 4 (4) | 2 (2) | 0 (0) | 0 (0)
lead insulation damage (Product Issues) | 2 (2) | 1 (1) | 4 (4) | 1 (1)
lead noise (Product Issues) | 4 (4) | 8 (8) | 8 (8) | 0 (0)
oversensing (Product Issues) | 3 (3) | 3 (3) | 4 (4) | 0 (0)
phrenic nerve/diaphragmatic stimulation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
shock due to AF with RVR (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
undersensing (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Durata Leads (N=982) | Riata Leads (N=670) | Riata ST Leads (N=458) | QuickSite/QuickFlex Leads (N=737)
Abnormal High Voltage Lead Impedance (Product Issues) | 2 (3) | 2 (2) | 0 (0) | 0 (0)
Abnormal Pacing Impedance (Product Issues) | 5 (6) | 1 (1) | 0 (0) | 3 (3)
Decrease R Wave (Product Issues) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Elevated pacing thresholds (Product Issues) | 3 (3) | 2 (2) | 1 (1) | 2 (2)
Lead Insulation Damage (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lead Noise (Product Issues) | 4 (4) | 1 (1) | 2 (2) | 0 (0)
Loss of Capture (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Loss of Sensing (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Other Visual Lead Anomalies (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Oversensing (Product Issues) | 4 (4) | 2 (2) | 3 (3) | 0 (0)
Oversensing Resulting in Therapy (Product Issues) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pectoral Stimulation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Phrenic Nerve/Diaphragmatic Stimulation (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Therapy for Non-Ventricular Rhythm (Product Issues) | 1 (1) | 3 (3) | 1 (1) | 0 (0)
Undersensing (Product Issues) | 0 (0) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review results communications prior to public release and embargo communications regarding trial results for 12 months from study completion date to allow time for multi-center study publication. After this period, the PI shall submit to sponsor for review a copy of any proposed manuscript at least 30 days prior to the estimated date of submission for publication. Sponsor may require delay of publication not to exceed 60 days for the purpose of filing patent applications.

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2015-09-18): https://cdn.clinicaltrials.gov/large-docs/87/NCT01507987/Prot_SAP_ICF_000.pdf